CLINICAL TRIAL: NCT00212173
Title: Behavioral & Pharmacologic Therapy of Adolescent Obesity
Brief Title: Adolescent Weight Management Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: DK54713 (completed 2007)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Protocol #1:Behavioral Therapy + Placebo or Sibutramine; Protocol #2: Behavioral Therapy + Meal Replacement or Conventional Food
Keywords: Adolescent; Weight Management; Obesity Treatment; Behavioral Treatment
MeSH Terms: interventions — sibutramine

INTERVENTIONS:
Drug: Sibutramine
Dietary Supplement: Slim Fast

SUMMARY:
Protocol #1:The goals of this study was to examine whether increased weight loss in obese adolescent is induced when the weight loss medication sibutramine is added to a family-based, behavioral weight control program.

Protocol #2: This study aims to improve the behavioral treatment of obesity during adolescence. A behavioral program using regular foods will be compared to a behavioral program using a structured meal plan (a portion-controlled approach with liquid-meal replacements [nutritional supplements]). This structured approach may be better for the promotion of weight loss compared to a diet of regular foods.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) between 28-50 kg/m2

Exclusion Criteria:

* Severe cardiovascular problems; arrhythmias
* Hypertension, uncontrolled (blood pressure >140/90 mm Hg)
* Diabetes mellitus (Fasting glucose > 126)
* Other serious medical disorders that would complicate dieting such as: Ulcer disease, cancer, thrombophlebitis, liver or kidney disease
* Current use of weight loss medications, amphetamines, steroids, or aspirin; medications affecting body weight
* Mental retardation or genetic syndromes associated with obesity
* Currently pregnant or planning a pregnancy or engaging in sexual activity without using contraceptives. All females will have a serum pregnancy test at baseline and all must agree to use contraception if they are sexually active during the study.
* Glaucoma
* History of major depression, bipolar disorder, or psychosis
* History of anorexia or bulimia
* Alcoholism and other substance abuse
* Use of anti-psychotic or anti-depressant medications in the last 6 months
* Highly dysfunctional family system or parental psychopathology
* Weight loss in the preceding 6 months of 5% or more and/or participation in another weight loss program
* Cigarette smoking or recent cessation
* If taking medication for hypertension or hypercholesterolemia condition must be stable for at least 3 months prior to enrollment in the study
* Chronic use of decongestants
* Intolerance of SlimFast

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120
Dates: Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Weight
BMI

SECONDARY OUTCOMES:
Blood Pressure
Lipids
Glucose
Insulin

CONTACTS AND LOCATIONS:
Overall Officials: Robert I Berkowitz, MD, Principal Investigator — Children's Hospital of Philadelphia

REFERENCES:
- [Result] Berkowitz RI, Wadden TA, Gehrman CA, Bishop-Gilyard CT, Moore RH, Womble LG, Cronquist JL, Trumpikas NL, Levitt Katz LE, Xanthopoulos MS. Meal replacements in the treatment of adolescent obesity: a randomized controlled trial. Obesity (Silver Spring). 2011 Jun;19(6):1193-9. doi: 10.1038/oby.2010.288. Epub 2010 Dec 9. PMID 21151016
- [Result] Bishop-Gilyard CT, Berkowitz RI, Wadden TA, Gehrman CA, Cronquist JL, Moore RH. Weight reduction in obese adolescents with and without binge eating. Obesity (Silver Spring). 2011 May;19(5):982-7. doi: 10.1038/oby.2010.249. Epub 2010 Oct 14. PMID 20948512